CLINICAL TRIAL: NCT00495131
Title: Randomized Trial of 24 or 48 Weeks of Peginterferon Alfa-2a Plus Ribavirin for Chronic Hepatitis C Virus Genotype 1-infected Patients in Taiwan
Brief Title: Randomized Trial of 24 or 48 Weeks of Peginterferon Alfa-2a Plus Ribavirin for HCV Genotype 1-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Dr. Jia-Horng Kao, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200705080M
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Genotype 1; Interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginterfron and ribavirin (24 weeks) (Active Comparator): Pegylated interferon alfa-2a (Pegasys, F. Hoffmann-LaRoche) 180 ug/week plus ribavirin (Robatrol, F. Hoffmann-LaRoche) 1000-1200 mg/day (<75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) for 24 weeks
  Interventions: Drug: Pegylated interferon alfa-2a plus ribavirin
- Peginterferon and ribavirin (48 weeks) (Active Comparator): Pegylated interferon alfa-2a (Pegasys, F. Hoffmann-LaRoche) 180 ug/week plus ribavirin (Robatrol, F. Hoffmann-LaRoche) 1000-1200 mg/day (<75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) for 48 weeks
  Interventions: Drug: Pegylated interferon alfa-2a plus ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a plus ribavirin — Pegylated interferon alfa-2a (Pegasys, F. Hoffmann-LaRoche) 180 ug/week plus ribavirin (Robatrol, F. Hoffmann-LaRoche) 1000-1200 mg/day (<75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) for 24 weeks
  Other Names: Pegasys plus Robatrol
  Arms: Peginterfron and ribavirin (24 weeks)
Drug: Pegylated interferon alfa-2a plus ribavirin — Pegylated interferon alfa-2a (Pegasys, F. Hoffmann-LaRoche) 180 ug/week plus ribavirin (Robatrol, F. Hoffmann-LaRoche) 1000-1200 mg/day (<75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) for 48 weeks
  Other Names: Pegasys plus Robatrol
  Arms: Peginterferon and ribavirin (48 weeks)

SUMMARY:
Chronic hepatitis C virus (HCV) infection is prevalent in the world, affecting 3% of the world's population. The current standard of therapy is pegylated interferon and ribavirin, reaching 54-63% of successful rates. In patients with HCV genotype 1 infection, a 48 week course of combination therapy has achieved a higher successful rate that a 24 weeks course of therapy. However, several studies in Taiwan have shown that a 24 week course of therapy has comparable or even better response to a 48 week course of therapy in Western countries. Therefore, whether a 48 week course of therapy can achieve a higher response to a 24 week course of therapy in Taiwanese patients with genotype 1 HCV infection remains unclear.

DETAILED DESCRIPTION:
Combination therapy with interferon alfa (IFN-α) plus ribavirin for 24 to 48 weeks produces sustained virologic response (SVR) rate in approximately 31-47% of treatment naïve patients with chronic hepatitis C.(1-5) Patients with genotype 1 virus infection are less likely to have SVR that those with other genotypes infection, and therefore, patients infected with hepatitis C virus (HCV) genotype 1 should receive treatment for 48 weeks.(6) Recently, combination therapy with pegylated interferon alfa (pegylated IFN-α) plus ribavirin produces higher SVR rates (54-56%) than that with IFN-α plus ribavirin.(7,8) Furthermore, a large trial assessing the effect and duration of pegylated IFN-α plus ribavirin showed that the overall SVR rate was 63%. Among patients with genotype 1 HCV infection, standard dose ribavirin (1000 to 1200 mg per day) and 48 weeks of treatment were significantly more effective than low dose ribavirin (800 mg per day) or 24 weeks of treatment.(9) The SVR rate was 51% for genotype 1 patients receiving pegylated IFN-α plus standard dose ribavirin for 48 weeks, whereas only 29% and 41% for those receiving pegylated IFN-α plus low dose ribavirin and standard dose ribavirin for 24 weeks, respectively. Based on these lines of evidence, 48 weeks of therapy with pegylated IFN-α (pegylated IFN-α 2a 180 μg or pegylated IFN-α 2b 1.5 μg per kilogram body weight weekly) plus ribavirin (1000 to 1200 mg per day) is recommended to treat patients with HCV genotype 1 infection.(10) In Taiwan, a multicenter study showed that a 6 month course treatment with pegylated IFN-α plus standard dose ribavirin had a comparable SVR rate to that with IFN-α plus standard dose ribavirin (67.1% versus 63.6%) in patients with chronic hepatitis C. Subgroup analysis showed that treatment with pegylated IFN-α plus standard dose ribavirin had a significantly higher SVR rate to that with IFN-α plus standard dose ribavirin (65.8% versus 41.0%) in patients with genotype 1 HCV infection.(11) Recently, a pilot study comparing 24 and 48 weeks of pegylated IFN-α plus standard dose ribavirin in patients with genotype 1 HCV infection showed that 48 weeks of treatment is more efficacious that 24 weeks of treatment (SVR rate: 80.0% versus 48.9%).(12) However, much difference of SVR rates occurred in these two studies, making optimal therapy in Taiwanese patients infected with genotype 1 HCV difficult to be determined. In the study, we aim to investigate in a large cohort whether 48 weeks treatment with pegylated IFN-α plus standard dose ribavirin is more efficacious than 24 weeks treatment in patients with genotype 1 HCV infection.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Age 18 and older than 18 years old
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Amplicor HCV Monitor v2.0, Roche Molecular Systems, Pleasanton, CA) with dynamic range 600~<500,000 IU/ml
* HCV genotype 1 (Inno-LiPA HCV II, Innogenetics, Ghent, Belgium)
* Serum alanine aminotransferase levels above the upper limit of normal with 6 months of enrollment
* A liver biopsy consistent with the diagnosis of chronic hepatitis C

Exclusion Criteria:

* Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
* Neutropenia (neutrophil count <1,500 per cubic milliliter)
* Thrombocytopenia (platelet <90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic alcohol abuse (daily consumption > 20 gram per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, MD, PhD, Study Chair — National Taiwan University Hospital; Ding-Shinn Chen, MD, Study Director — National Taiwan University Hospital; Ming-Yang Lai, MD, PhD, Study Director — National Taiwan University Hospital; Pei-Jer Chen, MD, PhD, Study Director — National Taiwan University Hospital; Chun-Jen Liu, MD, PhD, Principal Investigator — National Taiwan University Hospital; Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hosptial, Yun-Lin Branch; Chih-Lin Lin, MD, Principal Investigator — Ren-Ai Branch, Taipei City Hospital; Cheng-Chao Liang, MD, Principal Investigator — Far Eastern Memorial Hospital; Ching-Sheng Hsu, MD, Principal Investigator — Buddhist Tzu Chi General Hospital; Sheng-Shun Yang, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (6):
- Taiwan (6):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Buddhist Tzu Chi General Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Ren-Ai Branch, Taipei Municipal Hospital, Taipei

REFERENCES:
- [Background] McHutchison JG, Gordon SC, Schiff ER, Shiffman ML, Lee WM, Rustgi VK, Goodman ZD, Ling MH, Cort S, Albrecht JK. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. N Engl J Med. 1998 Nov 19;339(21):1485-92. doi: 10.1056/NEJM199811193392101. PMID 9819446
- [Background] Poynard T, Marcellin P, Lee SS, Niederau C, Minuk GS, Ideo G, Bain V, Heathcote J, Zeuzem S, Trepo C, Albrecht J. Randomised trial of interferon alpha2b plus ribavirin for 48 weeks or for 24 weeks versus interferon alpha2b plus placebo for 48 weeks for treatment of chronic infection with hepatitis C virus. International Hepatitis Interventional Therapy Group (IHIT). Lancet. 1998 Oct 31;352(9138):1426-32. doi: 10.1016/s0140-6736(98)07124-4. PMID 9807989
- [Background] Lai MY, Kao JH, Yang PM, Wang JT, Chen PJ, Chan KW, Chu JS, Chen DS. Long-term efficacy of ribavirin plus interferon alfa in the treatment of chronic hepatitis C. Gastroenterology. 1996 Nov;111(5):1307-12. doi: 10.1053/gast.1996.v111.pm8898645.
- [Background] Chemello L, Cavalletto L, Bernardinello E, Guido M, Pontisso P, Alberti A. The effect of interferon alfa and ribavirin combination therapy in naive patients with chronic hepatitis C. J Hepatol. 1995;23 Suppl 2:8-12. PMID 8720287
- [Background] Reichard O, Norkrans G, Fryden A, Braconier JH, Sonnerborg A, Weiland O. Randomised, double-blind, placebo-controlled trial of interferon alpha-2b with and without ribavirin for chronic hepatitis C. The Swedish Study Group. Lancet. 1998 Jan 10;351(9096):83-7. doi: 10.1016/s0140-6736(97)06088-1. PMID 9439491
- [Background] EASL International Consensus Conference on Hepatitis C. Paris, 26-28, February 1999, Consensus Statement. European Association for the Study of the Liver. J Hepatol. 1999 May;30(5):956-61. No abstract available. PMID 10365827
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] National Institutes of Health. National Institutes of Health Consensus Development Conference Statement: Management of hepatitis C: 2002--June 10-12, 2002. Hepatology. 2002 Nov;36(5 Suppl 1):S3-20. doi: 10.1053/jhep.2002.37117. No abstract available. PMID 12407572
- [Background] Lee SD, Yu ML, Cheng PN, Lai MY, Chao YC, Hwang SJ, Chang WY, Chang TT, Hsieh TY, Liu CJ, Chen DS. Comparison of a 6-month course peginterferon alpha-2b plus ribavirin and interferon alpha-2b plus ribavirin in treating Chinese patients with chronic hepatitis C in Taiwan. J Viral Hepat. 2005 May;12(3):283-91. doi: 10.1111/j.1365-2893.2005.00590.x. PMID 15850469
- [Background] Yu ML, Dai CY, Lin ZY, Lee LP, Hou NJ, Hsieh MY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL. A randomized trial of 24- vs. 48-week courses of PEG interferon alpha-2b plus ribavirin for genotype-1b-infected chronic hepatitis C patients: a pilot study in Taiwan. Liver Int. 2006 Feb;26(1):73-81. doi: 10.1111/j.1478-3231.2005.01196.x. PMID 16420512
- [Derived] Liu CH, Liu CJ, Lin CL, Liang CC, Hsu SJ, Yang SS, Hsu CS, Tseng TC, Wang CC, Lai MY, Chen JH, Chen PJ, Chen DS, Kao JH. Pegylated interferon-alpha-2a plus ribavirin for treatment-naive Asian patients with hepatitis C virus genotype 1 infection: a multicenter, randomized controlled trial. Clin Infect Dis. 2008 Nov 15;47(10):1260-9. doi: 10.1086/592579. PMID 18834319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 2006 June to September Location: academic centers
Pre-assignment Details: No wash out period in the study; all were treatment-naive All the patients who were eligible in the study were assigned to either groups without exclusion.
Groups:
- Peginterferon and Ribavirin (24 Weeks): Pegylated interferon alfa-2a (Pegasys, F. Hoffmann-LaRoche) 180 ug/week plus ribavirin (Robatrol, F. Hoffmann-LaRoche) 1000-1200 mg/day (<75 kg, 1000 mg/day; >= 75 kg, 1200 mg/day) for 24 weeks
Period: Overall Study
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks)
Started | 154 | 154
Completed | 147 | 148
Not Completed | 7 | 6
Not completed — Adverse Event | 6 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks) | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 128 | 250
  >=65 years | 32 | 26 | 58
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (10) | 53 (11) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 67 | 133
  Male | 88 | 87 | 175
Region of Enrollment [Number; unit: participants]
  Taiwan | 154 | 154 | 308

OUTCOME MEASURES:

1. Secondary Outcome: Treatment-related Withdrawal Rate
Description: Treatment-related withdrawal rate: patients who prematurely discontinued treatment due to treatment-related adverse events
Time Frame: 18 months
Measure: Number; unit: Participants
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks)
Number analyzed (Participants) | 154 | 154
Participants | 6 | 14

2. Primary Outcome: Sustained Virologic Response
Description: Undetectable HCV RNA 6 months off therapy
Time Frame: 18 months
Population: Intention-to-treat (ITT) analysis by last observation carried forward
Measure: Number; unit: participants
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks)
Number analyzed (Participants) | 154 | 154
participants | 87 | 117
Statistical Analysis 1: Comparison: Peginterferon and Ribavirin (24 Weeks) vs Peginterferon and Ribavirin (48 Weeks); Null hypothesis: no difference between 2 groups SVR estimation: 24 weeks (60%), 48 weeks (75%) alfa erros: 0.05, power: 0.80; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Primary Outcome: Sustained Biochemical Response
Description: Sustained biochemical response (SBR): alanine aminotransferase (ALT) normalization
Time Frame: 18 months
Population: Patients with end of follow-up alanine aminotransferase (ALT) levels
Measure: Number; unit: Participants
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks)
Number analyzed (Participants) | 147 | 148
Participants | 75 | 107

4. Secondary Outcome: Histologic Response
Description: Histologic response: improvement of at least 2 grade of scores by Ishak liver histologic classification by end of follow up liver biopsy to baseline liver biopsy
Time Frame: 18 months
Population: Data included for analysis only for patients with paired liver biopsies.
Measure: Number; unit: Participants
Arm/Group | Peginterferon and Ribavirin (24 Weeks) | Peginterferon and Ribavirin (48 Weeks)
Number analyzed (Participants) | 120 | 124
Participants | 71 | 97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No